CLINICAL TRIAL: NCT01278368
Title: PREOPERATIVE CHEMOTHERAPY DOES NOT ADVERSELY AFFECT SHORT-TERM OUTCOME AFTER PANCREATIC RESECTION.
Brief Title: Effect Of Preoperative Chemotherapy On Short-Term Outcome After Pancreatic Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Braga, Associate Professor of Surgery, Università Vita-Salute San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOADJUVANT_MATCH
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: pancreatic cancer, neoadjuvant chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preoperative chemotherapy (PCHT) (Active Comparator): Patients who underwent pancreatic resection after PCHT.
  Interventions: Procedure: Pancreatic resection after preoperative chemotherapy
- Control (Active Comparator): Patient who underwent pancreatic resection without preoperative therapy
  Interventions: Procedure: Pancreatic resection

INTERVENTIONS:
Procedure: Pancreatic resection after preoperative chemotherapy — Pancreatic resection after preoperative chemotherapy
  Arms: Preoperative chemotherapy (PCHT)
Procedure: Pancreatic resection — Pancreatic resection
  Arms: Control

SUMMARY:
No comparative trial investigating the effect of preoperative chemotherapy for locally advanced pancreatic cancer on short-term postoperative outcome has been published so far. The aim of the present study is to assess the potential impact of preoperative chemotherapy on short-term postoperative outcome after pancreatic resection in a case-matched series of cancer patients.

DETAILED DESCRIPTION:
Between 2003 and 2011, patients with locally advanced (stage III) pancreatic cancer who were treated with preoperative chemotherapy (PCHT) underwent surgical resection. Each patient was matched with the closest two patients with pancreatic cancer ( control group ) selected from our prospective electronic database who met the following match criteria: age (+/- 3 years), gender, ASA score, type of resection, pancreatic duct diameter (+/- 1 mm), and tumour size (+/- 5 mm).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatic cancer
* Preoperative chemotherapy
* Pancreatic resection

Exclusion Criteria:

* Metastatic disease
* ASA score 4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity rate | Postoperative. From 0 to 30 days after discharge

SECONDARY OUTCOMES:
Postoperative mortality | Postoperative. From 0 to 30 days after discharge
Length of hospital stay (LOS) | Postoperative. From 0 to 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marco Braga, MD, Principal Investigator — Università Vita-Salute San Raffaele
Locations (1):
- San Raffaele Hospital, Milan, Milan, Italy